CLINICAL TRIAL: NCT02342080
Title: Effects of System Suspended Robotic Lokomat Gait in Patients With Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0718.0.015.000-11
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Spinal Cord Injury
Keywords: Rehabilitation; Walking; Robotics; Neuronal Plasticity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional group (Experimental): A group with spinal cord injury will be trained in a 30-minute session 5 times weekly for 6 weeks. Each session will be supervised by qualified staff. Patients will undergo training with gradual increase in load and speed, according to the tolerance of each patient. The body weight support progression will start at 50 % of the patient body weight. It will be changed every 2 weeks and the load will decrease 10%. The progression of speed may be accompanied during the training period. For the robot locomotion therapy, the Lokomat system (Hocoma AG Switzerland) will be used.
  Interventions: Other: Training sessions; Device: Lokomat system (Hocoma AG Switzerland)

INTERVENTIONS:
Other: Training sessions — A group with spinal cord injury will be trained in a 30-minute session 5 times weekly for 6 weeks. Each session will be supervised by qualified staff. Patients will undergo training with gradual increase in load and speed, according to the tolerance of each patient. The body weight support progression will start at 50 % of the patient body weight. It will be changed every 2 weeks and the load will decrease 10%. The progression of speed may be accompanied during the training period.
Device: Lokomat system (Hocoma AG Switzerland) — For the robot locomotion therapy, the Lokomat system (Hocoma AG Switzerland) will be used.

SUMMARY:
Patients with incomplete spinal cord injury

DETAILED DESCRIPTION:
The objective of this project is to verify the effects of suspended robotic gait training (Lokomat) in recovery of functional capacity of the lower limbs patients with incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of incomplete spinal cord injury of traumatic origin
* Injury time from 1 to 36 months
* Stability verified in clinical medical evaluation
* ASIA C or D
* Absence of severe psychiatric amendment requiring psychiatric evaluations
* Present functional recovery of the upper limb compatible with stages III and IV of Brunnstrom
* Patients cannot use a cardiac pacemaker ; have unstable angina or other decompensated heart disease; have chronic obstructive pulmonary disease; dysreflexia without having autonomic control; have some fracture of the bones of the lower limbs; tracheostomy; presenting deformity and stiffness of the hip joint, knee (20 ° or more of flexion ) and ankle ( 10 or more plantar flexion ) and pressure ulcers.
* Absence of illicit drug use
* Grant writing the informed consent to participate in the study

Exclusion Criteria:

* Lack of resistance
* Disabling fatigue
* Worsening of spasticity which prevents the movement
* Body weight in excess of 150Kg
* Risk of osteoporosis with pathological fracture
* Asymmetry in the lower limbs greater than 2 cm
* Skin lesions and / or pressure ulcers in areas where the orthosis Lokomat pressuring

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Walking Index for Spinal Cord Injury II | 6 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linamara Rizzo Battistella, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Centro de Pesquisa Clínica do Instituto de Medicina Física e Reabilitação do HCFMUSP, São Paulo, São Paulo, Brazil